CLINICAL TRIAL: NCT07029347
Title: Correlation Hip Muscle Strength Of Dominant-Non-Dominant With Static Balance Parameters Using Stabilometry In Elderly Patients In Nursing Homes
Brief Title: Correlation Hip Muscle Strength With Static Balance Parameters In Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Irma Ruslina Defi, Principal Investigator, Universitas Padjadjaran
Other Study IDs: IKFR.11_1.06.25
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Geriatrics Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Strength of the dominant and non-dominant hip muscles using hydraulic pusj pull dynamometer — fleksor, ekstensor, abductor, adductor, internal rotasi, eksternal rotasi
Device: Static balance parameters using stabilometry — Center of Pressure (COP) range sway, velocity sway, dan weight distribution

SUMMARY:
Observational study aimed to identify the correlation between dominant and non-dominant hip muscle strength with static balance parameters using stabilometry (center of pressure (COP) range sway, velocity sway, and weight distribution) in elderly in nursing homes.

DETAILED DESCRIPTION:
24 elderly patients in nursing homes with an age range of 60-94 years were assessed using the Time Up and Go Test, Mini Mental State Exam (MMSE), Berg Balance Scale, 10 meter walking test, Activities-Specific Balance Confidence Scale, stabilometry and International Physical Activity Questionnaire (IPAQ) assessments as well as hip muscle strength examinations.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and above
* Able to walk indoors and outdoors without assistive devices
* Able to maintain a standing posture for 5 minutes without assistive devices
* Falls Efficacy Scale score below 20
* Time Up and Go test less than 13.5 seconds
* Able to read and write Latin letters
* Able to see images and writing on a television screen from a distance of 20 inches at 3 meters
* Able to understand exercise instructions (Mini Mental State Exam score ≥24/30 Indonesian version

Exclusion Criteria:

* Has a condition of high blood pressure (systolic >180 mmHg, heart rate at rest >120 bpm, blood glucose (GDS) >250 mg/dl), has symptoms of typical angina chest pain, shortness of breath, and severe headache
* Participants have undergone routine balance training within the last 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study used secondary data consisting of 24 participants from the Nursing Home. The gender of the participants was evenly divided, namely 12 men and 12 women. The age of the participants ranged from 60 - 94 years.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Strength of the dominant and non-dominant hip muscles | 6 weeks
  Strength of the dominant and non-dominant hip muscles using hydraulic push-pull dynamometer
Static balance parameters | 6 weeks
  Static balance parameters using stabilometry

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Sadikin General Hospital, Bandung, Indonesia

IPD SHARING:
Plan to Share IPD: No